CLINICAL TRIAL: NCT02101918
Title: Perfusion CT as Predictive Biomarker in a Phase II Study of Ziv-Aflibercept in Patients With Advanced Pancreatic Neuroendocrine Tumors
Brief Title: Ziv-Aflibercept in Treating and Computed Tomography Perfusion Imaging in Predicting Response in Patients With Pancreatic Neuroendocrine Tumors That Are Metastatic or Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-00642; NCI-2014-00642 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013-0954; 9604 (Other: M D Anderson Cancer Center); 9604 (Other: CTEP); N01CM00039 (NIH); P30CA016672 (NIH)
Record Dates: First submitted 2014-03-28; First posted 2014-04-02 (Estimated); Results first posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Multiple Endocrine Neoplasia Type 1; Pancreatic Neuroendocrine Carcinoma
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1; Somatostatinoma | interventions — Cytidine Triphosphate; aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (ziv-aflibercept, perfusion CT) (Experimental): Patients receive ziv-aflibercept IV over 60-120 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography perfusion imaging at baseline, day 21 of course 1, and at time of progression.
  Interventions: Radiation: Computed Tomography Perfusion Imaging; Other: Laboratory Biomarker Analysis; Biological: Ziv-Aflibercept

INTERVENTIONS:
Radiation: Computed Tomography Perfusion Imaging — Undergo computed tomography perfusion imaging
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Ziv-Aflibercept — Given IV
  Other Names: AFLIBERCEPT; AVE0005; Eylea; vascular endothelial growth factor trap; VEGF Trap; VEGF Trap R1R2; VEGF-Trap; Zaltrap

SUMMARY:
This phase II trial studies ziv-aflibercept in treating and perfusion computed tomography perfusion imaging in predicting response in patients with pancreatic neuroendocrine tumors that have spread to other parts of the body or cannot be removed by surgery. Ziv-aflibercept may stop the growth of tumor cells by blocking blood flow to the tumor. Diagnostic procedures, such as computed tomography perfusion, imaging may help measure a patient's response to ziv-aflibercept treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate the objective response rate (RR) of ziv-aflibercept among patients with advanced pancreatic neuroendocrine tumors (NET)s according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

II. Test the following hypotheses: that baseline perfusion computed tomography (CT) parameters can predict which patients with advanced pancreatic neuroendocrine tumors (pNETs) will respond to treatment with ziv-aflibercept.

SECONDARY OBJECTIVES:

I. Estimate progression free survival (PFS) duration among patients treated with ziv-aflibercept.

II. Evaluate the relationship between response rate and baseline blood volume (BV) and between response rate and baseline permeability surface (PS).

TERTIARY OBJECTIVES:

I. Determine whether post-treatment changes in BV expressed as relative change from baseline correlate with response to ziv-aflibercept.

II. Determine whether post-treatment tumor blood flow (BF) (absolute measurement) correlates with response to ziv-aflibercept.

III. Determine whether post-treatment changes in BF and, BV, expressed as relative change from baseline, correlate with relative change in sum of tumor diameters (RECIST 1.1 measurements).

IV. Determine the effect of ziv-aflibercept therapy on post-treatment blood flow (BF), BV, mean transit time (MTT), and PS at 4 weeks after treatment.

V. Evaluate the changes in tumor perfusion parameters at time of progression.

OUTLINE:

Patients receive ziv-aflibercept intravenously (IV) over 60-120 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography perfusion imaging at baseline, day 21 of course 1, and at time of progression.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed low or intermediate grade pancreatic NET; patients with neuroendocrine tumors associated with multiple endocrine neoplasia type 1 (MEN1) syndrome will be eligible
* Patients must have unresectable or metastatic disease
* Patients must have at least one measurable site of disease according to RECIST 1.1 that has not been previously irradiated
* Patients must have at least one lesion suitable for perfusion CT; the lesion should be greater than or equal to 3 cm in size in the cranial caudal direction
* Patient must have no contraindication for CT with iodinated contrast
* Patients who are on a somatostatin analogue for control of hormonal syndromes must be on a stable dose (no change in mg dose of long acting octreotide or lanreotide, changes in dosing interval of +/- 1 week is allowed) for 2 months prior to date of study entry
* Women of child-bearing potential must have a negative serum pregnancy test within 7 days prior to date of study entry; women who have had menses within the past 2 years, who have not had a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy are considered to be of child-bearing potential; patients with elevated human chorionic gonadotropin (hCG) at baseline that is judged to be related to the tumor are eligible if hCG levels do not show the expected doubling when repeated 5-7 days later, or pregnancy has been ruled out by vaginal ultrasound
* Any number of prior lines of systemic anti-neoplastic therapy are allowed; treatment with =< 1 prior VEGF inhibitor will be allowed
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Urine protein:creatinine ratio =< 1.0 OR 24-hour urine protein =< 500 mg (24-hour total urine protein only need be obtained if urine protein:creatinine ratio < 1.0)
* Patients must have prothrombin time (PT)/international normalized ratio (INR)/partial thromboplastin time (PTT) within 1.2 x the upper limit of normal
* Patients must have resting blood pressure (BP) no greater than 140 mmHg (systolic) or 90 mmHg (diastolic) for eligibility; initiation or adjustment of BP medication is permitted prior to study entry
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Less than 28 days elapsed from prior radiotherapy, from prior surgery and prior chemotherapy to the time of randomization; less than 42 days elapsed from prior major surgery to the time of randomization
* Adverse events (with exception of alopecia, peripheral sensory neuropathy and those listed in specific exclusion criteria) from any prior anti cancer therapy of grade > 1 (National Cancer Institute Common Terminology Criteria [NCI CTCAE] version [v.]4.0)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) > 2
* History of brain metastases, uncontrolled spinal cord compression, or carcinomatous meningitis or new evidence of brain or leptomeningeal disease
* Other prior malignancy; adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix or any other cancer from which the patient has been disease free for > 5 years are allowed
* Participation in another clinical trial and any concurrent treatment with any investigational drug within 30 days prior to study entry
* Any of the following within 6 months prior to study entry: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association (NYHA) class III or IV congestive heart failure, stroke or transient ischemic attack
* Any of the following within 3 months prior to study entry: grade 3-4 gastrointestinal bleeding/hemorrhage, treatment resistant peptic ulcer disease, erosive esophagitis or gastritis, infectious or inflammatory bowel disease, diverticulitis, pulmonary embolism or other uncontrolled thromboembolic event
* Occurrence of deep vein thrombosis within 4 weeks, prior to study entry
* Acquired immuno deficiency syndrome (AIDS-related illnesses) or known human immunodeficiency virus (HIV) disease requiring antiretroviral treatment
* Any severe acute or chronic medical condition, which could impair the ability of the patient to participate to the study or to interfere with interpretation of study results
* Pregnant or breast feeding women; positive pregnancy test (serum or urine beta-human chorionic gonadotropin [HCG]) for women of reproductive potential
* Patient with reproductive potential (female and male) who do not agree to use an accepted effective method of contraception (hormonal or barrier methods, abstinence) during the study treatment period and for at least 3 months following completion of study treatment; for female patient enrolled, the following methods of contraception are acceptable: oral contraceptives accompanied by the use of a second method of contraception, or intra uterine device (IUD) or women who are surgically sterile, or women who are post -menopausal or other reasons have no chance of becoming pregnant
* Absence of signed and dated Institutional Review Board-approved patient informed consent from prior to enrollment in the study
* EXCLUSION CRITERIA RELATED TO ZIV-AFLIBERCEPT
* Urine protein-creatinine ratio (UPCR) > 1 urinalysis or total urine protein > 500 mg/24 hours (h)
* Serum creatinine > 1.5 x upper limit of normal (ULN); if creatinine 1.0-1.5 x ULN, creatinine clearance, calculated according to Cockcroft-Gault formula, < 60 ml/min will exclude the patient
* History of uncontrolled hypertension, defined as systolic blood pressure > 150 mmHg while simultaneous diastolic blood pressure > 100 mmHg, or systolic blood pressure > 180 mmHg when diastolic blood pressure < 90 mmHg, on at least 2 repeated determinations on separate days within 3 months prior to study enrollment
* Patients on anticoagulant therapy with unstable dose of warfarin and/or having an out-of- therapeutic range INR (> 3) within the 4 weeks prior to study entry
* Evidence of clinically significant bleeding diathesis or underlying coagulopathy (e.g. INR > 1.5 without vitamin K antagonist therapy), non-healing wound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-06-18 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Halperin, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - M D Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Aflibercept 6 mg /kg IV: Aflibercept 6 mg /kg IV every 3 weeks.
Period: Overall Study
Arm/Group | Aflibercept 6 mg /kg IV
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Aflibercept 6 mg /kg IV
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 5
Age, Continuous [Mean (Full Range); unit: years] | 60.3 [36 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate According to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Description: 90% exact confidence interval was constructed for the overall group. Per Response EvaluationCriteria In SolidTumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR)=CR+PR,
Time Frame: Through study completion an average of 19 months
Population: Eligible patients with baseline perfusion CT imaging. One patient from moffitt was a screen fail however 21 patients were evaluable for response and toxicity.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Aflibercept 6 mg /kg IV
Number analyzed (Participants) | 21
percentage of participants | 9.5 [1.7 to 27.1]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Calculated for all eligible participants using the Kaplan Meier method and reported with confidence interval.
Time Frame: Through study completion an average of 19 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Aflibercept 6 mg /kg IV
Number analyzed (Participants) | 21
months | 10.4 [1.97 to 17.73]

3. Secondary Outcome: Baseline Blood Volume (BV)
Description: The relationship between response rate and baseline BV will be evaluated. In addition to hypothesis testing using externally generated cut-points, refinement of optimal cut points in baseline BV separating responders and non-responders will be performed. Receiver operating characteristic (ROC) curves will be generated. Response rates of perfusion computed tomography (pCT) subgroups defined by these cut-points will be compared using chi-square test. Response profiles of pCT subgroups defined by these cut-points will be compared using non-parametric test (Wilcoxon rank sum test).
Time Frame: Baseline
Population: Due to low response rate data were not collected
Arm/Group | Aflibercept 6 mg /kg IV
Number analyzed (Participants) | 0

4. Secondary Outcome: Baseline Permeability Surface (PS)
Description: The relationship between response rate and baseline PS will be evaluated. In addition to hypothesis testing using externally generated cut-points, refinement of optimal cut points in baseline PS separating responders and non-responders will be performed. ROC curves will be generated. Response rates of pCT subgroups defined by these cut-points will be compared using chi-square test. Response profiles of pCT subgroups defined by these cut-points will be compared using non-parametric test (Wilcoxon rank sum test).
Time Frame: Baseline
Population: Due to low response rate data were not collected
Arm/Group | Aflibercept 6 mg /kg IV
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Change in BV
Description: Median will be used as cut point for correlation of post-treatment changes in BV expressed as relative change from baseline with response. Response rates will be compared using chi-square test or Fisher's exact test whenever appropriate. Response profiles will be compared using non-parametric test (Wilcoxon rank sum test).
Time Frame: Baseline to 4 weeks after treatment
Population: Due to the low response rate, data for blood volume were not collected
Arm/Group | Aflibercept 6 mg /kg IV
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Post-treatment Tumor Blood Flow (BF)
Description: Median will be used as cut point for correlation of post-treatment tumor BF (absolute measurement) with response. Response rates will be compared using chi-square test or Fisher's exact test whenever appropriate. Response rates will be compared using chi-square test or Fisher's exact test whenever appropriate.
Time Frame: 4 weeks after treatment
Population: Response rate was too low to power a valid analysis.
Arm/Group | Aflibercept 6 mg /kg IV
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Post-treatment Change in BF
Description: Continuous parameters in relative change in pCT parameters will be plotted against best relative change in sum of tumor diameters from RECIST 1.1 tumor measurements. Pearson correlation will be used to test statistical significance. Non-parametric test will be used if appropriate.
Time Frame: Baseline to 4 weeks after treatment
Population: Response rate was too low to power a valid analysis.
Arm/Group | Aflibercept 6 mg /kg IV
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Post-treatment Change in BV
Description: as for outcome 7
Time Frame: Baseline to 4 weeks after treatment
Population: Response rate was too low to power a valid analysis.
Arm/Group | Aflibercept 6 mg /kg IV
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Change in Participants Parameters
Description: The effect of ziv-aflibercept therapy on post-treatment BF, BV, mean transit time, and PS will be determined. Descriptive statistics of pre and post treatment values will be given. Distribution of pre and post treatment values will be graphed. Treatment induced change in values will be compared using paired-t test. Non-parametric test will be used if appropriate.
Time Frame: Baseline to 4 weeks after treatment
Population: Response rate was too low to power a valid analysis.
Arm/Group | Aflibercept 6 mg /kg IV
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: Tumor Perfusion Parameters at Time of Progression
Time Frame: Up to 1 year
Population: No patients underwent perfusion CT at time of progression, no analysis could not be performed.
Arm/Group | Aflibercept 6 mg /kg IV
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: C1D1 and for 30 days after the last dose of study drug.
Description: Patients will be followed until resolution or stabilization of the adverse event.
Arm/Group | Aflibercept 6 mg /kg IV
All-Cause Mortality (participants affected / at risk) | 1/22
Serious Adverse Events (participants affected / at risk) | 4/22
Other Adverse Events (participants affected / at risk) | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aflibercept 6 mg /kg IV (N=22)
Pain Abdominal (Gastrointestinal disorders) | 1
Hemorrhage Upper GI (Blood and lymphatic system disorders) | 1
cholecystitis (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aflibercept 6 mg /kg IV (N=22)
Abdominal pain (Gastrointestinal disorders) | 5
Alanine aminotransferase increased (Investigations) | 4
Anemia (Blood and lymphatic system disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Aspartate aminotransferase increased (Investigations) | 3
Constipation (Gastrointestinal disorders) | 5
Creatinine increased (Investigations) | 3
Diarrhea (Gastrointestinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Fatigue (General disorders) | 6
Headache (Nervous system disorders) | 15
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 9
Hypertension (Vascular disorders) | 17
Mucositis oral (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 5
Neutrophil count decreased (Investigations) | 3
Pain (General disorders) | 3
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3
Platelet count decreased (Blood and lymphatic system disorders) | 3
Proteinuria (Renal and urinary disorders) | 7
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Weight loss (Metabolism and nutrition disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/18/NCT02101918/Prot_SAP_000.pdf